CLINICAL TRIAL: NCT01077375
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Switch Study to Evaluate the Safety, Tolerability and Efficacy of Milnacipran in Patients With an Inadequate Response to Duloxetine for the Treatment of Fibromyalgia
Brief Title: Study of Milnacipran in Patients With Inadequate Response to Duloxetine for the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Cypress Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN-MD-28
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Results first posted 2012-01-26 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2011-12

CONDITIONS: Fibromyalgia
Keywords: Milnacipran; Duloxetine; Switch; Forest Research Institute
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablets, twice a day, oral administration
  Interventions: Drug: Placebo
- Milnacipran (Experimental): Milnacipran tablets, 100 to 200 mg/day, oral administration, twice daily in divided doses.
  Interventions: Drug: Milnacipran

INTERVENTIONS:
Drug: Placebo — * Placebo tablets, oral administration, twice daily for 10 weeks during randomized, double-blind treatment period. Duloxetine capsules, oral administration, 30 mg/day for 1 week after randomization to effect a duloxetine down-taper.
  * Placebo tablets, twice daily for 1 week during double-blind down-taper treatment period.
  Arms: Placebo
Drug: Milnacipran — * Milnacipran tablets, 100 to 200 mg/day, oral administration, twice daily in divided doses for 10 weeks during randomized, double-blind treatment period. Placebo capsules, 1 capsule/day administered for 1 week after randomization to maintain double-blind duloxetine down-taper.
  * Milnacipran tablets, 100 to 0 mg/day, oral administration, twice daily in divided doses for 1 week during double-blind down-taper treatment period.
  Other Names: Savella
  Arms: Milnacipran

SUMMARY:
The objective of this study is to evaluate the safety, tolerability and efficacy of milnacipran in patients with an inadequate response to duloxetine for the treatment of fibromyalgia.

DETAILED DESCRIPTION:
* Two weeks Duloxetine 60 mg Open-Label Period
* Randomization to Double-Blind Treatment Period: 10 weeks Milnacipran (direct switch) or 10 weeks placebo (one week blinded 30 mg duloxetine)
* One week Double-Blind Down-Taper Period

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia
* Have been treated with a stable dosage of duloxetine (60 mg/day) for ≥ 4 weeks immediately before Screening (Visit 1)
* Duloxetine must have been prescribed for the treatment of Fibromyalgia
* Have a VAS 1-week pain recall score ≥ 40 mm and ≤ 90 mm
* At Visit 2, to be eligible to enter the randomized treatment period, must continue to have a VAS 1-week pain recall score ≥ 40 mm and be dissatisfied with current Duloxetine treatment.

Exclusion Criteria:

* Suicidal risk
* History of mania, bipolar disorder, psychotic disorder, schizophrenia, or a current episode of major depressive disorder
* Myocardial infarction and/or stroke within the prior 6 months
* Systolic blood pressure > 160 mm Hg or mean diastolic blood pressure > 100 mm Hg at Screening (Visit 1)
* Substance abuse
* Pulmonary dysfunction
* Severe renal impairment
* Active cardiac disease
* Liver disease
* Uncontrolled narrow-angle glaucoma
* Autoimmune disease
* Cancer
* Inflammatory bowel disease
* Unstable endocrine disease
* Prostatic enlargement
* Female patients who are pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Spera, Study Director — Forest Research Institute Inc., A Subsidiary of Forest Laboratories
Locations (26):
- United States (26):
  - Forest Investigative Site 013, Sacramento, California
  - Forest Investigative Site 022, Cromwell, Connecticut
  - Forest Investigative Site 021, Danbury, Connecticut
  - Forest Investigative Site 007, Delray Beach, Florida
  - Forest Investigative Site 008, Ocala, Florida
  - Forest Investigative Site 009, Orlando, Florida
  - Forest Investigative Site 016, Orlando, Florida
  - Forest Investigative Site 012, St. Petersburg, Florida
  - Forest Investigative Site 019, Tampa, Florida
  - Forest Investigative Site 006, Atlanta, Georgia
  - Forest Investigative Site 024, Atlanta, Georgia
  - Forest Investigative Site 015, Evansville, Indiana
  - Forest Investigative Site 005, Worchester, Massachusetts
  - Forest Investigative Site 010, Jackson, Mississippi
  - Forest Investigative Site 025, St Louis, Missouri
  - Forest Investigative Site 018, Willingboro, New Jersey
  - Forest Investigative Site 014, Syracuse, New York
  - Forest Investigative Site 023, Charlotte, North Carolina
  - Forest Investigative Site 002, Cincinnati, Ohio
  - Forest Investigative Site 003, Cleveland, Ohio
  - Forest Investigative Site 001, Medford, Oregon
  - Forest Investigative Site 020, Mechanicsburg, Pennsylvania
  - Forest Investigative Site 011, Greer, South Carolina
  - Forest Investigative Site 004, Salt Lake City, Utah
  - Forest Investigative Site 017, Bellevue, Washington
  - Forest Investigative Site 026, Racine, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred over an 8 month period from February 2010 to September 2010 at 25 study centers in the United States. Last patient last visit occurred on December 22nd, 2010.
Pre-assignment Details: All participants were given an open-label treatment of duloxetine 60 mg once daily for a two week period before randomization.
  Patients randomized to placebo received 1 week of duloxetine 30 mg to effect a duloxetine down-taper. Patients randomized to milnacipran received 1 week of placebo capsules to maintain the blind.
Groups:
- Placebo: Randomized Population: placebo treatment assignment, dose-matched placebo tablets, twice a day, oral administration.
- Milnacipran: Randomized Population: milnacipran treatment assignment, 100 to 200 mg/day, twice a day in divided doses, oral administration.
Period: Overall Study
Arm/Group | Placebo | Milnacipran
Started | 21 | 86 (One randomized patient not taking study drug was excluded from the Double-blind Safety Population.)
Completed | 11 | 51
Not Completed | 10 | 35
Not completed — Adverse Event | 2 | 15
Not completed — Lack of Efficacy | 6 | 8
Not completed — Withdrawal by Subject | 0 | 6
Not completed — Lost to Follow-up | 2 | 5
Not completed — Other Reason | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Double-blind Safety Population: Placebo treatment assignment, dose-matched placebo tablets, twice a day, oral administration.
- Milnacipran: Double-blind Safety Population: milnacipran treatment assignment, 100 to 200 md/day, twice a day in divided doses, oral administration.
  One patient randomized to the milnacipran treatment group did not take at least one dose of double-blind study drug and was therefore not included in the Double-blind Safety Population.
- Total: Total of all reporting groups
Arm/Group | Placebo | Milnacipran | Total
Number analyzed (Participants) | 21 | 85 | 106
Age Continuous [Mean (Standard Deviation); unit: years] | 48.5 (11.3) | 48.5 (10.5) | 48.5 (10.6)
Age, Customized [Number; unit: participants]
  18 to 59 | 17 | 77 | 94
  60 to 70 | 4 | 8 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 79 | 98
  Male | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 21 | 85 | 106

OUTCOME MEASURES:

1. Primary Outcome: Responder Status Based on Patient Global Impression of Change (PGIC) Score at Visit 5 (Week 13)
Description: The PGIC is a patient-reported measure of improvement in pain sensation and quality of life scored on a scale from 1 (very much improved) to 7 (very much worse). To meet the criteria for a responder in this study, patients must report a score of 1 (very much improved) or 2 (much improved) on the PGIC.
Time Frame: Assessed at Visit 4 (Week 9) and Visit 5 (Week 13) or early termination. Presented results generated via LOCF approach.
Population: ITT Population: patients in the Double-blind Safety Population with ≥ 1 PGIC post-baseline assessment. Double-blind Safety Population includes 6 patients who were not included in ITT population. Presented results generated via LOCF approach. No statistical comparisons between groups are presented; study was exploratory, not hypothesis-testing.
Measure: Number; unit: participants
Groups:
- Placebo: Intent-to-treat (ITT) Population, placebo treatment assignment, dose-matched placebo tablets, twice a day, oral administration.
- Milnacipran: Intent-to-treat Population, milnacipran treatment assignment, 100 to 200 mg/day, twice a day, oral administration.
  Flexible dosing from 50 mg/day to 200 mg/day was allowed except at a) the initial dosage after randomization had to be 100 mg/day, b) the dose range during week 1 of the randomized double-blind treatment period was 50 to 100 mg/day, and c) patients had to be on at least 100 mg/day at Visit 3 (Week 5).
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 21 | 79
participants | 5 | 26

2. Secondary Outcome: Change From Baseline to Visit 5 (Week 13) in the Visual Analog Scale (VAS) 1-week Pain Recall Score
Description: The VAS assessment ranges from a scale of 0 (no pain) to 100 (worst possible pain).
Time Frame: Change from Baseline (Week 3) to Visit 5 (Week 13)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Placebo: Intent-to-treat Population, placebo treatment assignment, dose-matched placebo tablets, twice a day, oral administration.
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 21 | 79
Units on a scale | -1.3 (22.5) | -12.3 (27.3)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a nearly 10 month period from March 4th, 2010 through December 22, 2010.
Groups:
- Milnacipran: Double-blind Safety Population: milnacipran treatment assignment, 100 to 200 mg/day, twice a day, oral administration.
  One patient randomized to the milnacipran treatment group did not take at least one dose of double-blind study drug and was therefore not included in the Double-blind Safety Population.
  Flexible dosing from 50 mg/day to 200 mg/day was allowed except at a) the initial dosage after randomization had to be 100 mg/day, b) the dose range during week 1 of the randomized double-blind treatment period was 50 to 100 mg/day, and c) patients had to be on at least 100 mg/day at Visit 3 (Week 5).
Arm/Group | Placebo | Milnacipran
Serious Adverse Events (participants affected / at risk) | 0/21 | 2/85
Other Adverse Events (participants affected / at risk) | 16/21 | 63/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Milnacipran (N=85)
Hypersensitivity (Immune system disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Milnacipran (N=85)
Nausea (Gastrointestinal disorders) | 6 | 18
Dizziness (Nervous system disorders) | 1 | 13
Headache (Nervous system disorders) | 2 | 10
Insomnia (Psychiatric disorders) | 2 | 9
Hot flush (Vascular disorders) | 1 | 7
Irritability (General disorders) | 1 | 6
Nasopharyngitis (Infections and infestations) | 0 | 6
Anxiety (Psychiatric disorders) | 0 | 5
Blood pressure increased (Investigations) | 0 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 5
Diarrhea (Gastrointestinal disorders) | 3 | 4
Fatigue (General disorders) | 2 | 3
Migraine (Nervous system disorders) | 2 | 1
Paresthesia (Nervous system disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.